CLINICAL TRIAL: NCT03458325
Title: Economic Impact of Reducing Hospital Admissions for Patients Presenting to the Emergency Department With Worsening Heart Failure: An Adaptive Clinical Trial of Furoscix Infusor
Brief Title: Furoscix Real-World Evaluation for Decreasing Hospital Admissions in Heart Failure
Acronym: FREEDOM-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: scP-01-005
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: A prospective treatment arm (i.e., Furoscix administered via the Furoscix Infusor) administered outside the hospital that will be compared to a propensity-matched historical control arm of patients admitted to the hospital for ≤ 72 hours (i.e., Treatment As Usual (TAU)) that will be derived from administrative claims data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Furoscix Infusor Prospective Treatment (Experimental): Furoscix (furosemide injection, 8 mg/mL) administered subcutaneously over 5 hours via the Furoscix Infusor outside the hospital.
  Interventions: Combination Product: Furoscix Infusor
- Propensity-Matched Historical Control (No Intervention): The control arm will be populated with claims data for patients with HF and fluid overload who presented to the emergency department and were admitted to the hospital for ≤ 72 hours for the treatment of HF with intravenous diuretics. Patients admitted for diuresis-only will be identified by using diagnostic codes for admittance from a claims database.

INTERVENTIONS:
Combination Product: Furoscix Infusor — Furoscix Infusor, a drug-device combination product for subcutaneous delivery of Furoscix, buffered furosemide injection, 8 mg/mL (total dose = 80 mg dose) administered subcutaneously for 5 hours.
  Arms: Furoscix Infusor Prospective Treatment

SUMMARY:
The study is to evaluate the safe admission avoidance and the overall economic impact associated with management of worsening HF using the drug-device combination product, the Furoscix Infusor, outside the hospital setting in patients initially presenting to the emergency department.

The study drug, Furoscix (furosemide injection 8 mg/ml), is a furosemide solution buffered to a neutral pH containing 80 mg/10 mL for subcutaneous administration over 5 hours via the Furoscix Infusor.

The study objectives are:

1. To evaluate differences in healthcare resource utilization and direct medical costs for patients treated with the Furoscix Infusor outside the hospital versus patients receiving intravenous furosemide for ≤ 72 hours in the hospital setting for 30 days post-discharge from the emergency department.
2. To evaluate the safety of Furoscix administered outside the hospital.
3. To evaluate and describe quality of life and patient satisfaction for patients who receive the Furoscix Infusor outside the hospital setting.

DETAILED DESCRIPTION:
This adaptive clinical trial will include a prospective treatment arm (i.e., Furoscix administered via the Furoscix Infusor) administered outside the hospital that will be compared to a propensity-matched historical control arm of patients admitted to the hospital for ≤ 72 hours (i.e., Treatment As Usual (TAU)) that will be derived from administrative claims data. Eligible patients for the Furoscix arm will be patients with HF and fluid overload who initially present to the emergency department (ED) and who are expected to require parenteral diuresis.

If it is determined by the investigator that the patient requires parenteral diuresis or continued diuresis outside of the ED care setting and meets all study eligibility criteria, he/she may be consented and enrolled into the study.

The treatment comprises a preprogrammed bi-phasic 5-hour drug administration. Subjects will be instructed on the use of the Furoscix Infusor by the investigator and/or study staff in accordance with the instructions for use. The initial dose of the study product may be administered in the ED or at home. Additional doses will be provided to the subject for self-administration or administration by a caregiver in the home setting as directed by the investigator or study staff. The total duration in days and total number of doses of the initial therapy will be determined by the investigator based on an estimated volume of diuresis desired to transition patient back to their oral diuretic maintenance therapy. Subjects will receive scheduled at-home telephone calls from a HF nurse on Days 1 and 7 and one call between Days 14-21. Planned in-clinic visits will be conducted between Day 2-4 and then Day 30. Unscheduled at-home telephone calls by a HF nurse and unscheduled in-clinic visits may be performed if felt clinically indicated by the study team or the clinical provider.

The study period will be up to 30 days after enrollment. All outcomes will be assessed up to 30 days after the initial discharge from the emergency department.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. NYHA Class II-III HF presenting to the emergency department for worsening HF at baseline
3. On background therapy includes those receiving 40-160 mg of oral furosemide equivalents daily (20-80 mg Torsemide or 1-4 mg Bumetanide).
4. Signs of extracellular volume expansion, defined as one or more of the following:

   1. jugular venous distention
   2. pitting edema (≥1+),
   3. abdominal distension
   4. pulmonary congestion on chest x-ray
   5. pulmonary rales
5. After initial emergency department evaluation and treatment (i.e., at the time of the care transition decision*), candidates for parenteral diuresis outside of the hospital, defined as all the following:

   1. Oxygen saturation ≥ 90% on exertion
   2. Respiratory Rate < 24 breaths per minute
   3. Resting Heart Rate < 100 beats per minute
   4. Systolic Blood Pressure > 100 mmHg
6. Adequate environment for at-home administration of Furoscix

Exclusion Criteria:

1. Presence of a complicating condition, other than HF that requires immediate hospitalization or anticipated hospitalization in the next 30 days
2. Evidence of acute renal failure as determined at the discretion of the investigator
3. Known allergy to the active and inactive ingredients of the study medication or device adhesive
4. Any local abdominal skin condition on the day of treatment i.e. sunburn, rash, eczema, etc.
5. Currently participating in another interventional research study
6. Women who are pregnant or who could become pregnant and are not willing to use an adequate form of contraception
7. Estimated Creatinine Clearance < 30 mL per minute by Cockcroft-Gault equation

   CrCl (mL/min) = {(140 - age) x Lean Body Weight (kg)/Serum Creatinine (mg/dL) x 72} (x 0.85 if female)
8. If baseline creatinine value is available: an increase of ≥ 0.5 mg/dL in creatinine from baseline
9. HF requiring immediate hospitalization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Olive View - UCLA Medical Center, Sylmar, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Ascension St. Vincent Heart Center, Indianapolis, Indiana
  - Unity Point Health, Des Moines, Iowa
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Abington Hospital - Jefferson Health, Abington, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects excluded after signing consent:
  * 1 subject met exclusion criteria due to lab abnormality (creatinine clearance, serum creatinine)
  * 1 subject met exclusion criteria due to requiring hospitalization (hypoxia and hypertension)
Period: Overall Study
Arm/Group | Furoscix Infusor Prospective Treatment
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Subject's Insurance at baseline [Count of Participants; unit: Participants]
  Medicare | 8
  Medicaid | 4
  Commercial | 10
  Unknown | 2
NYHA Classification [Count of Participants; unit: Participants] — New York Heart Association Classification
  * Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea.
  * Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  * Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  * Class IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest that worsen with physical activity.
  Participants
    NYHA Class I | 0
    NYHA Class II | 4
    NYHA Class III | 20
    NYHA Class IV | 0
Signs of volume expansion at baseline [Count of Participants; unit: Participants]
  Jugular Venous Distention | 4
  Pitting Edema | 18
  Abdominal Distention | 9
  Pulmonary Congestion on Chest X-ray | 6
  Pulmonary Rales | 5
History of Congestive Heart Failure (CHF) [Mean (Standard Deviation); unit: Years] | 4.26 (4.917)
Etiology of Congestive Heart Failure (CHF) at baseline [Count of Participants; unit: Participants]
  Ischemic | 9
  Non-ischemic | 15

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Utilization Costs
Description: The difference in the overall and heart failure related healthcare costs between subjects treated with the Furoscix Infusor through 30 days post discharge from the emergency department compared to matched controls treated in the hospital for ≤ 72 hours through 30 days post discharge.
Time Frame: Day 0 - Day 30
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
US Dollars
  HF-related healthcare costs | 2920.30 (7073.20)
  Overall healthcare costs | 7512.30 (11,905.50)
Statistical Analysis 1: Comparison: Furoscix Infusor Prospective Treatment; The comparator arm was populated with claims data for patients who presented to the emergency department for worsening HF and were admitted to the hospital for ≤ 72 hours for the treatment of HF. The filter was further strengthened by analyzing diagnostic codes and resource utilization during their hospital stay to exclude hospitalizations other than Heart Failure. Each subject from the Furoscix group was matched to controls in ratios ranging from 1:1 to 4:1; Test type: Superiority; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -16,995.30, 95% CI 2-sided [-22,187.90 to -11,802.70]

2. Secondary Outcome: Heart-Failure Related Hospital Admissions
Description: The HF-related admissions for the Furoscix patients compared to Control patients.
Time Frame: Day 0 - Day 30
Population: Evaluable Population:
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
Participants | 1
Statistical Analysis 1: Comparison: Furoscix Infusor Prospective Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6765, Fisher Exact; Percentage Difference = -6.4

3. Secondary Outcome: All-Cause Hospital Admissions
Description: The differences in the percentage of subjects with an all-cause hospitalization in the Furoscix group and all-cause 30-day rehospitalization in the Control group in the 30 day follow-up period
Time Frame: Day 0 - Day 30
Population: Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
Participants | 6
Statistical Analysis 1: Comparison: Furoscix Infusor Prospective Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5856, Fisher Exact; Mean Difference (Net) = 5.3

4. Secondary Outcome: Heart-Failure Related Emergency Department Visits
Description: The differences in the percentage of patients with HF-related emergency department visits in the Furoscix group and in the Control group in the 30 day follow-up period
Time Frame: Day 0 - Day 30
Population: Evaluable Population
Measure: Count of Participants; unit: Participants
Groups:
- Matched Historical Control: The control arm was populated with claims data for patients who presented to the emergency department for worsening HF and were admitted to the hospital for ≤ 72 hours for the treatment of HF.
Arm/Group | Furoscix Infusor Prospective Treatment | Matched Historical Control
Number analyzed (Participants) | 24 | 66
Participants | 1 | 4
Statistical Analysis 1: Comparison: Furoscix Infusor Prospective Treatment vs Matched Historical Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.000, Fisher Exact; Mean Difference (Net) = -1.9

5. Secondary Outcome: Heart-Failure Related Clinic Visits
Description: The differences in the percentage of patients with HF-related clinic visits in the Furoscix group and in the Control group in the 30 day follow-up period
Time Frame: Day 0 - Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
Participants | 24
Statistical Analysis 1: Comparison: Furoscix Infusor Prospective Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Chi-squared; Mean Difference (Net) = 65.1

6. Secondary Outcome: KCCQ-12 Scores
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) measures a patient's self-reported overall health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life (QOL). The KCCQ-12 overall summary score is the sum of responses from all 12 items ranging from 0 to 100 with higher scores to indicate better health status.
Time Frame: 30 Days
Population: Summary Score represents integration of Physical Limitation, Symptom Frequency, Quality of Life and Social Limitation Scores. Missing values were not included in this analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Furoscix Infusor Prospective Treatment - Baseline; Furoscix Infusor Prospective Treatment - Day 30: Furoscix (furosemide injection, 8 mg/mL) administered subcutaneously over 5 hours via the Furoscix Infusor outside the hospital.
  Furoscix Infusor: Furoscix Infusor, a drug-device combination product for subcutaneous delivery of Furoscix, buffered furosemide injection, 8 mg/mL (total dose = 80 mg dose) administered subcutaneously for 5 hours.
Arm/Group | Furoscix Infusor Prospective Treatment - Baseline | Furoscix Infusor Prospective Treatment - Day 30
Number analyzed (Participants) | 24 | 24
score on a scale
  Summary Score: number analyzed (Participants) | 21 | 21
  Summary Score | 29.9 (22.8) | 42.8 (28.4)
  Physical Limitation Score: number analyzed (Participants) | 23 | 23
  Physical Limitation Score | 37.1 (30.1) | 43.7 (32.0)
  Symptom Frequency Score | 33.1 (28.6) | 50.5 (32.3)
  Quality of Life Score | 27.1 (28.0) | 35.9 (29.8)
  Social Limitation Score: number analyzed (Participants) | 22 | 22
  Social Limitation Score | 29.0 (26.1) | 40.9 (31.3)
Statistical Analysis 1: Comparison: Furoscix Infusor Prospective Treatment - Baseline vs Furoscix Infusor Prospective Treatment - Day 30; Analysis for Summary Score; Test type: Superiority; p = 0.0443, t-test, 2 sided; P-value was obtained from the paired t-test statistic; Mean Difference (Net) = 12.8, 95% CI 2-sided [0.4 to 25.3]

7. Secondary Outcome: Mean Change in NT-proBNP and BNP
Description: Change in NT-proBNP and BNP change from baseline during the study period is summarized for the Furoscix group
Time Frame: Day 0 - Day 30
Population: Evaluable Population. Subjects who are missing the NT-proBNP and BNP test results were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Furoscix Infusor Prospective Treatment - Baseline | Furoscix Infusor Prospective Treatment - Day 30
Number analyzed (Participants) | 23 | 23
pg/ml
  NT-proBNP: number analyzed (Participants) | 11 | 10
  NT-proBNP | 823.4 (1043.9) | 700.7 (896.2)
  BNP: number analyzed (Participants) | 12 | 13
  BNP | 785.1 (1129.9) | 263.5 (384.0)
Statistical Analysis 1: Comparison: Furoscix Infusor Prospective Treatment - Baseline vs Furoscix Infusor Prospective Treatment - Day 30; Test type: Superiority — Statistical Analysis for the mean change in NT-proBNP over 30 days; p = 0.5133, t-test, 2 sided; Mean Difference (Final Values) = -122.6, 95% CI 2-sided [-525.8 to 280.5]
Statistical Analysis 2: Comparison: Furoscix Infusor Prospective Treatment - Baseline vs Furoscix Infusor Prospective Treatment - Day 30; Statistical Analysis for mean change in BNP over 30 days; Test type: Superiority; p = 0.0420, t-test, 2 sided; Mean Difference (Final Values) = -719.9, 95% CI 2-sided [-1406.5 to -33.2]

8. Secondary Outcome: Comfort of Wear Questionnaire
Description: The Furoscix group was administered a Comfort of Wear Questionnaire during Day 2-4 study visit. This questionnaire measured the patient's general perception of comfortability wearing and using the device, the impact of wearing the device on their activities of daily living, and their satisfaction with the device.
Time Frame: Day 0 - Day 2-4 study visit
Population: Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
Participants
  Please rate how comfortable or uncomfortable you felt wearing the device: Very Comfortable | 6
  Please rate how comfortable or uncomfortable you felt wearing the device: Moderately Comfortable | 9
  Please rate how comfortable or uncomfortable you felt wearing the device: Slightly Comfortable | 3
  Please rate how comfortable or uncomfortable you felt wearing the device: Neither Comfortable or Uncomfortable | 0
  Please rate how comfortable or uncomfortable you felt wearing the device: Slightly Uncomfortable | 5
  Please rate how comfortable or uncomfortable you felt wearing the device: Moderately Uncomfortable | 1
  Please rate how comfortable or uncomfortable you felt wearing the device: Very Uncomfortable | 0
  Please rate how comfortable or uncomfortable you felt upon removal of the device: Very Comfortable | 11
  Please rate how comfortable or uncomfortable you felt upon removal of the device: Moderately Comfortable | 4
  Please rate how comfortable or uncomfortable you felt upon removal of the device: Slightly Comfortable | 2
  Please rate how comfortable or uncomfortable you felt upon removal of the device: Neither Comfortable or Uncomfortable | 4
  Please rate how comfortable or uncomfortable you felt upon removal of the device: Slightly Uncomfortable | 1
  Please rate how comfortable or uncomfortable you felt upon removal of the device: Moderately Uncomfortable | 1
  Please rate how comfortable or uncomfortable you felt upon removal of the device: Very Uncomfortable | 1

9. Secondary Outcome: Comfort of Wear Questionnaire: Interference With Activities Daily Living
Description: The Furoscix group was administered a Comfort of Wear Questionnaire on Day 2-4. This questionnaire measured the patient's general perception of comfortability wearing and using the device, the impact of wearing the device on their activities of daily living, and their satisfaction with the device.
Time Frame: Day 0 - Day 2-4 study visit
Population: Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
Participants
  If wearing the device interfered with activities of daily living - Walking: 1 - Not at all | 19
  If wearing the device interfered with activities of daily living - Walking: 2 - Probably Not | 1
  If wearing the device interfered with activities of daily living - Walking: 3 - Possibly | 1
  If wearing the device interfered with activities of daily living - Walking: 4 - Probably | 1
  If wearing the device interfered with activities of daily living - Walking: 5 - Completely | 1
  If wearing the device interfered with activities of daily living - Walking: Not Applicable | 1
  If wearing the device interfered with activities of daily living - Standing: 1 - Not at all | 19
  If wearing the device interfered with activities of daily living - Standing: 2 - Probably Not | 1
  If wearing the device interfered with activities of daily living - Standing: 3 - Possibly | 1
  If wearing the device interfered with activities of daily living - Standing: 4 - Probably | 1
  If wearing the device interfered with activities of daily living - Standing: 5 - Completely | 1
  If wearing the device interfered with activities of daily living - Standing: Not Applicable | 1
  If wearing the device interfered with activities of daily living - Sitting reading watching TV: 1 - Not at all | 17
  If wearing the device interfered with activities of daily living - Sitting reading watching TV: 2 - Probably Not | 5
  If wearing the device interfered with activities of daily living - Sitting reading watching TV: 3 - Possibly | 0
  If wearing the device interfered with activities of daily living - Sitting reading watching TV: 4 - Probably | 0
  If wearing the device interfered with activities of daily living - Sitting reading watching TV: 5 - Completely | 1
  If wearing the device interfered with activities of daily living - Sitting reading watching TV: Not Applicable | 1
  If wearing the device interfered with activities of daily living - Lying down/napping: 1 - Not at all | 13
  If wearing the device interfered with activities of daily living - Lying down/napping: 2 - Probably Not | 4
  If wearing the device interfered with activities of daily living - Lying down/napping: 3 - Possibly | 2
  If wearing the device interfered with activities of daily living - Lying down/napping: 4 - Probably | 2
  If wearing the device interfered with activities of daily living - Lying down/napping: 5 - Completely | 0
  If wearing the device interfered with activities of daily living - Lying down/napping: Not Applicable | 3
  If wearing the device interfered with activities of daily living - Using the bathroom: 1 - Not at all | 17
  If wearing the device interfered with activities of daily living - Using the bathroom: 2 - Probably Not | 2
  If wearing the device interfered with activities of daily living - Using the bathroom: 3 - Possibly | 1
  If wearing the device interfered with activities of daily living - Using the bathroom: 4 - Probably | 3
  If wearing the device interfered with activities of daily living - Using the bathroom: 5 - Completely | 1
  If wearing the device interfered with activities of daily living - Using the bathroom: Not Applicable | 0
  If wearing the device interfered with activities of daily living - Driving or riding in a car: 1 - Not at all | 14
  If wearing the device interfered with activities of daily living - Driving or riding in a car: 2 - Probably Not | 4
  If wearing the device interfered with activities of daily living - Driving or riding in a car: 3 - Possibly | 1
  If wearing the device interfered with activities of daily living - Driving or riding in a car: 4 - Probably | 0
  If wearing the device interfered with activities of daily living - Driving or riding in a car: 5 - Completely | 0
  If wearing the device interfered with activities of daily living - Driving or riding in a car: Not Applicable | 5

10. Secondary Outcome: Comfort of Wear Questionnaire: Subject and/or Caregiver Satisfaction
Description: as for outcome 8
Time Frame: Day 0 - Day 2-4 study visit
Population: Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor Prospective Treatment
Number analyzed (Participants) | 24
Participants
  I think that I would like to use this product frequently: 1 - Strongly Disagree | 0
  I think that I would like to use this product frequently: 2 - Disagree | 2
  I think that I would like to use this product frequently: 3 - Neutral | 7
  I think that I would like to use this product frequently: 4 - Agree | 2
  I think that I would like to use this product frequently: 5 - Strongly Agree | 13
  I found the product unnecessarily complex: 1 - Strongly Disagree | 14
  I found the product unnecessarily complex: 2 - Disagree | 7
  I found the product unnecessarily complex: 3 - Neutral | 0
  I found the product unnecessarily complex: 4 - Agree | 1
  I found the product unnecessarily complex: 5 - Strongly Agree | 2
  I thought the product was easy to use: 1 - Strongly Disagree | 0
  I thought the product was easy to use: 2 - Disagree | 2
  I thought the product was easy to use: 3 - Neutral | 0
  I thought the product was easy to use: 4 - Agree | 4
  I thought the product was easy to use: 5 - Strongly Agree | 18
  I think that I would need the support of a technical person to be able to use this product: 1 - Strongly Disagree | 22
  I think that I would need the support of a technical person to be able to use this product: 2 - Disagree | 0
  I think that I would need the support of a technical person to be able to use this product: 3 - Neutral | 1
  I think that I would need the support of a technical person to be able to use this product: 4 - Agree | 0
  I think that I would need the support of a technical person to be able to use this product: 5 - Strongly Agree | 1
  I found the various functions in this product were well integrated: 1 - Strongly Disagree | 2
  I found the various functions in this product were well integrated: 2 - Disagree | 2
  I found the various functions in this product were well integrated: 3 - Neutral | 2
  I found the various functions in this product were well integrated: 4 - Agree | 4
  I found the various functions in this product were well integrated: 5 - Strongly Agree | 14
  I thought there was too much inconsistency in this product: 1 - Strongly Disagree | 18
  I thought there was too much inconsistency in this product: 2 - Disagree | 5
  I thought there was too much inconsistency in this product: 3 - Neutral | 1
  I thought there was too much inconsistency in this product: 4 - Agree | 0
  I thought there was too much inconsistency in this product: 5 - Strongly Agree | 0
  I would imagine that most people would learn to use this product very quickly: 1 - Strongly Disagree | 0
  I would imagine that most people would learn to use this product very quickly: 2 - Disagree | 0
  I would imagine that most people would learn to use this product very quickly: 3 - Neutral | 0
  I would imagine that most people would learn to use this product very quickly: 4 - Agree | 1
  I would imagine that most people would learn to use this product very quickly: 5 - Strongly Agree | 23
  I found the product very cumbersome to use: 1 - Strongly Disagree | 11
  I found the product very cumbersome to use: 2 - Disagree | 4
  I found the product very cumbersome to use: 3 - Neutral | 5
  I found the product very cumbersome to use: 4 - Agree | 1
  I found the product very cumbersome to use: 5 - Strongly Agree | 3
  I felt very confident using the product: 1 - Strongly Disagree | 0
  I felt very confident using the product: 2 - Disagree | 0
  I felt very confident using the product: 3 - Neutral | 0
  I felt very confident using the product: 4 - Agree | 5
  I felt very confident using the product: 5 - Strongly Agree | 19
  I needed to learn a lot of things before I could get going with this product: 1 - Strongly Disagree | 15
  I needed to learn a lot of things before I could get going with this product: 2 - Disagree | 3
  I needed to learn a lot of things before I could get going with this product: 3 - Neutral | 2
  I needed to learn a lot of things before I could get going with this product: 4 - Agree | 3
  I needed to learn a lot of things before I could get going with this product: 5 - Strongly Agree | 1

ADVERSE EVENTS:
Time Frame: 30 Days from Enrollment
Arm/Group | Furoscix Infusor Prospective Treatment
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 18/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Furoscix Infusor Prospective Treatment (N=24)
Cardiac Failure Congestive (Cardiac disorders) | 1
Food Poisoning (Gastrointestinal disorders) | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1
Hyperosmolar State (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Lymphedema (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Furoscix Infusor Prospective Treatment (N=24)
Infusion Site Hemorrhage (General disorders) | 2
Infusion Site Bruising (General disorders) | 7
Infusion Site Pain (General disorders) | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Urinary Tract Infection (Infections and infestations) | 2
Dizziness (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT03458325/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03458325/SAP_001.pdf